CLINICAL TRIAL: NCT06780592
Title: The Efficacy of Vebreltinib Combined With Temozolomide for Glioblastoma (GBM) After Surgery: a Study Protocol for a Prospective, Open-label ,Multi-center, Randomized, Controlled Trial in China
Brief Title: Vebreltinib Combined With Temozolomide for Glioblastoma (GBM) After Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-754
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
Keywords: Vebreltinib; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, randomized, open-label, clinical trial in China.
  The plan is to recruit 60 eligible subjects and assign them to either the control group (standard TMZ 5/28 therapy) or the experimental group (TMZ plus LEV Vebreltinib) at a 1:1 ratio. Participants will undergo a 48-week treatment period and a 2-year follow-up period.. The study is expected to commence recruitment in mainland China in about Aug 2024. It is expected that the trial will end in December 2025.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vebreltinib + Temozolomide (Experimental): Participants received Vebreltinib (300 mg Bid) in combination with Temozolomide (150 mg/m2) treatment, every 4 weeks for up to 6 cycles (Induction).
  Interventions: Drug: Vebreltinib + Temozolomide
- Temozolomide (Active Comparator): Participants received Temozolomide (150 mg/m2) treatment, every 4 weeks for up to 6 cycles (Induction).
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Vebreltinib + Temozolomide — Vebreltinib is a capsule in the form of 25 mg and 100mg, twice daily. Participants received Vebreltinib (300 mg Bid) in combination with Temozolomide (150 mg/ m2) treatment, every 4 weeks for up to 6 cycles (Induction).
  Arms: Vebreltinib + Temozolomide
Drug: Temozolomide — Participants received Temozolomide (150 mg/ m2) treatment, every 4 weeks for up to 6 cycles (Induction).
  Arms: Temozolomide

SUMMARY:
The purpose of this study is to explore the effects of Vebreltinib in primary glioblastoma patients receiving a combination therapy of chemotherapy (temozolomidel) and MET-TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years, female or male
2. Newly diagnosed GBM (WHO grade 4) patients with maximal surgical resection
3. c-MET overexpression diagnosed by IHC
4. KPS ≥60
5. Adequate hematological, renal, and hepatic function.

   All patients should meet the following criteria:
   1. absolute neutrophil count (ANC) ≥1.5 × 109/L and platelet count≥100 × 109/L
   2. serum creatinine clearance ≥80 mL/min
   3. total bilirubin level ≤ 1.5 × ULN (except patients with Gilbert syndrome)
   4. aspartate aminotransferase (AST) ≤ 3.0 × ULN, alanine aminotransferase (ALT) ≤ 3.0 × ULN, and AST/ALT < 2.5 × ULN
6. The patient and his/her family members were informed and provided signed and informed consent

Exclusion Criteria:

1. Any previous postoperative treatment except for concurrent chemoradiotherapy;
2. Individuals unable to undergo cranial MRI examination;
3. Active hemorrhage detected by cranial CT or MRI scan before enrollment;
4. Uncontrolled hypertension;
5. Decompensated heart failure, unstable angina pectoris, acute myocardial infarction, or persistent and clinically significant arrhythmias within 3 months before enrollment;
6. Anti-HIV (+), or both anti-HCV and HCV-RNA (+), or HBsAg positive with HBV-DNA >1000IU/ml;
7. Individuals requiring long-term continuous use of hematopoietic growth factors or platelet transfusions;
8. Pregnant or lactating women;
9. Individuals who have received other clinical trial drugs within 30 days before the first dose of the study drug;
10. Individuals deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Every 4 weeks (±14 days) from enrollment until the last enrolled participant completes a 12-month follow-up or is lost to follow-up.
  The primary outcome is the PFS of patients, the time from randomization and group allocation to any recorded disease progression, and even death.

SECONDARY OUTCOMES:
Overall survival (OS) | Every 4 weeks (±14 days) from enrollment until the last enrolled participant completes a 12-month follow-up or is lost to follow-up.
  The time from randomization and allocation to death for any reason
The Karnof sky Performance status scale (KPS) | Every 4 weeks (±14 days) from enrollment until the last enrolled participant completes a 12-month follow-up or is lost to follow-up.
  The scale measures the levels of patient activity and medical needs. The score ranges from 100 (no signs of disease) to 0 (dead).
Objective response rate (ORR) | Every 4 weeks (±14 days) from enrollment until the last enrolled participant completes a 12-month follow-up or is lost to follow-up.
  Objective response rate (ORR) = (CR + PR)/total number of cases × 100%. A complete response (CR) is defined as the disappearance of all target lesions. A partial response (PR) is defined as a reduction of at least 30% in the sum of diameters of the target lesions, considering the baseline sum diameters as a reference. The ORR will be determined by MRI according to the Response Evaluation Citeria in Solid Tumors (RECIST)
Incidence of adverse events (AEs) | Every 4 weeks (±14 days) from enrollment until the last enrolled participant completes a 12-month follow-up or is lost to follow-up.
  Adverse events (CTC-Toxicity ≥ grade III) will be recorded and analyzed based on the Common Terminology Criteria for Adverse Events (CTC-AE)

IPD SHARING:
Plan to Share IPD: No